CLINICAL TRIAL: NCT01182233
Title: Evaluation of a Method Designed to Improve Outcome of HD Chemotherapy and AHSCT for Patients With Myeloma: Total Marrow Irradiation Administered Via Helical Tomotherapy Plus High-Dose Melphalan and Amifostine Before AHSCT2
Brief Title: Total Skeletal Irradiation in Multiple Myeloma Before Second Autologous Hematopoietic Stem Cell Transplantation
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: low enrollment
Sponsor: University of Rochester (Other)
Responsible Party: Principal Investigator, Gordon Phillips, MD, Professor of Medicine, Division of Hematology/Oncology, University of Rochester
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 30850
Record Dates: First submitted 2010-08-03; First posted 2010-08-16 (Estimated); Last update posted 2016-05-17 (Estimated); Status verified 2015-04

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma; Autologous Hematopoietic Stem Cell Transplant; Total Skeletal Irradiation; High dose chemotherapy
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Total Skeletal Irradiation (Experimental): Three subjects determined to be eligible for study and agree to participate are assigned to receive 200 cGy of TSI-HT for 5 days. If this dose level is well tolerated in the first 3 subjects, the dose will be increased and given over 5 days. The dose will continue to be increased until the maximum toelrated dose is reached.
  Interventions: Radiation: Total Skeletal Irradiation

INTERVENTIONS:
Radiation: Total Skeletal Irradiation — Escalating doses of TSI starting at 200cGy (escalating up to 400cGy unless maximum tolerated dose is determined in lower dose level) in cohort 1 over 5 days followed by high dose melphalan and cytoprotection followed by autologous hematopoietic stem cell transplant

SUMMARY:
The purpose of this study is to improve the efficacy of the HDC regimen by adding a novel, "targeted" means administering a variation of total body irradiation (TBI) radiation i.e., total skeletal irradiation (TSI) administered by helical tomotherapy (HT) before, and in addition to the current standard of HDC, at a dose of 200 mg/m2 (HDMel200). The underlying postulate of this endeavor is that TSI-HT will provide additional cytoreduction to HDMel alone, without producing additional (serious) toxicity. We will utilize a classical Phase I study design (i.e., dose escalation) in myeloma patients undergoing AHSCT2 to define a maximum tolerated dose (MTD) and dose limiting toxicity (DLT). Finally, although comparisons to other therapies are not typical (and/or feasible) for a Phase I study, we will compare, whenever possible, both the toxicity and the antimyeloma activity of the AHSCT2 to AHSCT1.

This protocol will standardize, as much as possible the use of AHSCT2 both as a "tandem" and "salvage" procedure. Since sufficient AHSC (CD34+ cells) are routinely collected in adequate numbers for multiple AHSCTs, but recently used infrequently, it is important to work towards defining the optimal utilization of this resource.

DETAILED DESCRIPTION:
While HDC/AHSCT is active most patients eventually relapse; obviously, those with lesser responses progress as well. Many investigators regard HDC/AHSCT as a "mature" modality a useful if fixed element in an evolving treatment paradigm that focuses on the introduction of new (non-HDC/AHSCT) agents with unique mechanisms of action. However, data from several related sources (including both the syngeneic and second ["tandem" or salvage] AHSCT experience), suggests that the efficacy of HDC/AHSCT could be improved by obtaining better cytoreduction of the HDC component, thus prolonging survival and possibly even producing an increase in cures. However, to do so will require additional attention to the sources of relapse following HDC/AHSCT, mainly the residual myeloma in the patient, but perhaps also the inadvertent reinfusion of clonogenic myeloma cells in the AHSCT. For reasons discussed herein, this study will focus on the former.

We believe that the agents with more potent activity vs. the (multiple) myeloma cancer stem cell (MM-CSC) and/or their microenvironment are ultimately needed to increase the cure rate in myeloma. Unfortunately, preliminary data suggest current modalities used in myeloma therapy are only variably effective vs. these targets, and that newer agents with such activity are only now becoming available for clinical trials.

The use of these newer agents are most likely to augment, not supplant, current modalities, lending even more urgency to optimizing existing elements to try to improve the efficacy of HDC/AHSCT and especially to determine if activity vs. MM-CSC and/or the microenvironment of these current modalities can be augmented. Radiation seems especially attractive to re-evaluate, given new, "targeted" methods of administration such as those described herein. Impetus for this effort comes from the known radiosensitivity of clonogenic myeloma cells (a population that at least may contain MM-CSC), and especially given the ability of local radiotherapy to provide local disease control in myeloma, and especially given the ability of local radiotherapy to cure some patients with solitary plasmacytoma "proving" activity of radiotherapy vs. MM-CSC in this closely-related diagnosis.

It is important to note that improvement in current modalities may offer better clinical outcomes even if major effects vs. the MM-CSC and microenvironment interaction are not produced. We do not currently have the ability to measure such effects; this will not be part of this trial.

ELIGIBILITY:
Inclusion Criteria:

* Age </= 70 years
* Documented myeloma confirmed at protocol entry
* Adequate presence of >/=2.0x10e6/kg cryopreserved CD34+ cells
* Adequate organ function
* Prior therapy is allowed as long as the organ function parameters are maintained and/or excessive radiation exposure is not produced
* Chemosensitivity

Exclusion Criteria:

* Uncontrolled infection
* Pregnant or lactating females
* Patients in >/= very good partial response after initial primary non-transplant therapy and/or AHSCT1
* Patients unwilling to practice adequate forms of contraception if clinically indicated

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2010-06; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Define the maximum tolerated dose of a derived high dose therapy regimen | Day 100 post transplant
  MTD of high dose therapy consisting of escalating doses of Total Skeletal Irradiation administered via Helical Tomotherapy, followed by standard high dose chemotherapy of high dose Melphalan (200mg/m2) with amifostine cytoprotection before AHSCT.

SECONDARY OUTCOMES:
Determine the dose-limiting toxicity (DLT) of TSI-HT therapy | Day 100 post transplant
  This objective will also include detailed short and long term assessment of hematopoiesis even if it is not the dose limiting toxicity.
Compare toxicities to those produced by the AHSCT1 regimen | Day 100 post transplant
  Determine if quantity and severity of toxicities of TSI regimen are less than toxicities experienced in AHSCT1.
Compare antitumor results obtained by TSI-HT before AHSCT | End of study (June 2013 - anticipated)
  Compare using standard outcome parameters (ie; response rate, relapse rate, disease-free survival or progression-free survival and overall survival) to high dose chemotherapy/AHSCT1

CONTACTS AND LOCATIONS:
Overall Officials: Gordon Phillips, MD, Principal Investigator — University of Rochester
Locations (1):
- University of Rochester Medical Center, Rochester, New York, United States